CLINICAL TRIAL: NCT04385628
Title: The Factors Affecting the Emotional Reactions of Relatives of Intensive Care Patients to the News of Death.
Brief Title: Breaking the Bad News to the Bereaved Family and Their Reactions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Bülent Barış Güven, medical doctor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 48670771-514.10
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: The Effective Factors on the Grief Reactions to the Death Information
Keywords: patient death , grief reactions

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relatives of patients hospitalized in the intensive care unit: Demographic data of the relative of the patient (age, proximity, educational background, patient co-existence, ethnicity, marital status, number of children, history of psychological treatment and the presence of an intensive care treatment history of any family member before) will be recorded. After the 3rd, 10th, and 30th days of patient admission, and once a month, the patient satisfaction survey will be filled face to face during informing the patient's relative. These three main data (Demographic data of the patient relatives, the most recent satisfaction questionnaire and emotional reactions observed while reporting death) will be evaluated and interpreted.
  Interventions: Behavioral: the patient' relatives satisfaction questionnaire

INTERVENTIONS:
Behavioral: the patient' relatives satisfaction questionnaire — The patient' relatives satisfaction questionnaire will be filled face to face during informing the patient's relatives after the 3rd, 10th, and 30th days of patient admission, and once a month. We will evaluate the most recent questionnaire.

SUMMARY:
The demographic characteristics, satisfaction survey evaluations and emotional reactions of the relatives of the patients who are admitted to the intensive care unit and who have an expected mortality rate higher than 50% according to the Apache-2 scoring system will be investigated.

DETAILED DESCRIPTION:
Patients with an APACHE-2 score> 25 (Expected mortality rate> 50%) during the first 24 hours of hospitalization in the Intensive Care Unit will be included in the study. A person who comes to the most frequent visit from relatives of patients will be included in the study. Demographic data of the relative of the patient after the informed volunteer consent form has been approved (age, proximity, educational background, patient co-existence, ethnicity, marital status, number of children, history of psychological treatment and the presence of an intensive care treatment history of any family member before) will be registered. After the 3rd, 10th, and 30th days of patient admission, and once a month, the patient satisfaction survey will be filled face to face during informing the patient's relative. In this patient group with an expected mortality of> 50%, if death occurs, the information will be made to the visitor of the patient who frequently visits the patient and agrees to participate in the study. The emotional reaction of the relative of the patient participating in the study during the declaration of death will be recorded in the case report form.

Grief reaction is unique, and it will differ from one individual to another. Possible reactions of relatives of patients during the death notification (Emotional Reactions)

1. Regular response; In this case, the relatives of the patients often describe the event as expected or my patient is now free from suffering.
2. Initial shock reaction; It may be complete desperation and a state of closure,
3. Denial- This is an initial defense mechanism after the unexpected, devastating news, and it should be recognized and tolerated. Acceptance may be possible by encouraging the relatives to view the body of the deceased, especially to those relatives who were not present at the time of death
4. Anger- This is a common reaction after the sudden death of a beloved relative. The expression of this anger can vary from mild irritation to violent behavior. This can be expressed on self, hospital staff, or any other person. Anger will gradually diminish once expressed
5. Guilt- This is nothing but the inward expression of anger and self-blame. Consoling words of the health care team will help to do away with this emotion.

ELIGIBILITY:
Inclusion Criteria:

* Apache 2 score> 25 or Expected death rate> 50%,
* Hospitalization period> 72 hours in intensive care unit -

Exclusion Criteria:

* Apache 2 score <25 or Expected death rate <50%,
* Those who have a stay in ICU <72 hours
* Currently receiving psychological medication
* Those who do not accept one of the legal heirs to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Relatives of patients hospitalized in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-09-29 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Regular response to the bad news | From admission to discharge, up to 3 month
  These three main data (Demographic data of the patient relatives, the most recent satisfaction questionnaire and emotional reactions observed while reporting death) will be evaluated and interpreted.
Initial shock reactions to the bad news | From admission to discharge, up to 3 month
  These three main data (Demographic data of the patient relatives, the most recent
Denial to the bad news | From admission to discharge, up to 3 month
  These three main data (Demographic data of the patient relatives, the most recent
Anger to the bad news | From admission to discharge, up to 3 month
  These three main data (Demographic data of the patient relatives, the most recent
Guilt to the bad news | From admission to discharge, up to 3 month
  These three main data (Demographic data of the patient relatives, the most recent

CONTACTS AND LOCATIONS:
Overall Officials: selçuk Taşçı, Study Chair — Sultan Abdulhamidhan Training Hospital; ayşın ersoy, Study Director — Sultan Abdulhamidhan Training Hospital
Locations (1):
- Sultan 2.Abdulhamidhan training hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Naik SB. Death in the hospital: Breaking the bad news to the bereaved family. Indian J Crit Care Med. 2013 May;17(3):178-81. doi: 10.4103/0972-5229.117067. PMID 24082616
- [Result] Jurkovich GJ, Pierce B, Pananen L, Rivara FP. Giving bad news: the family perspective. J Trauma. 2000 May;48(5):865-70; discussion 870-3. doi: 10.1097/00005373-200005000-00009. PMID 10823529